CLINICAL TRIAL: NCT00138944
Title: Effectiveness of Eplerenone to Improve Target Organ Damage in Patients With Resistant Arterial Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Roland E. Schmieder, Prof. Dr. med., University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFO_TP5/2; DFG KFO 106-2 TP5
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- 2 (Active Comparator): Eplerenone
  Interventions: Drug: eplerenone

INTERVENTIONS:
Drug: placebo — od
  Arms: 1
Drug: eplerenone — 50mg od
  Arms: 2

SUMMARY:
Resistant hypertension is defined as hypertension not controlled (i.e. blood pressure not below 140/90 mmHg) with the use of adequate doses of at least three different anti-hypertensives including a diuretic. Resistant hypertension is abundant. In the ALLHAT trial 34% of patients did not reach the blood pressure goal of 140/90 mmHg. One possible mechanism of resistance is the aldosterone-escape phenomenon.

During aldosterone escape, aldosterone plasma levels are normal or even elevated despite therapy with ACEIs or ARBs. The prevalence is about 30-50%. Possible reasons for aldosterone escape are alternative ways of aldosterone stimulation (hyperkalemia, adrenomedullin, ACTH), local aldosterone production or primary aldosteronism. Aldosterone has deleterious blood pressure independent effects on cardiac, vascular and renal damage.

Hypothesis: Eplerenone is effective to improve hypertensive target organ damage in patients with resistant hypertension.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Casual blood pressure >=140/90 despite effective triple therapy including an ACEI/ARB and a diuretic

Exclusion Criteria:

* Contraindication for eplerenone
* Creatinine-Clearance < 60 ml/min
* Diabetes mellitus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Change of left ventricular mass | 3 months vs. baseline
  MRT assessment of left ventricular mass

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, MD, Study Chair — University Erlangen-Nuremberg
Locations (1):
- CRC Medical Department IV, Erlangen, Germany